Can Vitamin D Reduce Heart Muscle Damage After Bypass Surgery?

NCT04323852

24/10/2020

## Statistical analysis:

The patients' number (35 patients per group) was determined based on the previous trials investigating the caspase activity in the CABG setting.15,22,23 Categorical variables were reported as numbers and percentages, whereas mean + standard deviation was expressed for continuous variables. Repeated measures of analysis of variance and multiple comparisons were applied using the Bonferroni correction (type I error correction), to evaluate the change of measured inflammatory markers between the groups by over time. The Kolmogorov-Smirnov test was performed for normality. Continuous variables and categorical variables were compared between groups using Student t test (or Mann-Whitney test for those meeting abnormal distribution) and w2, respectively. All the statistical analyses were performed using SPSS version 23 (SPSS, Chicago, Illinois). A P value <.05 was considered as significant.